CLINICAL TRIAL: NCT02189187
Title: Keeping Weight Off: Brain Changes Associated With Healthy Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Carl Fulwiler, Associate Professor of Psychiatry, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R34AT006963 (NIH)
Record Dates: First submitted 2014-06-24; First posted 2014-07-14 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Overweight; Obesity
Keywords: Weight Loss; Body Weight Changes; Body Weight; Magnetic Resonance Imaging; Emotions; Emotion regulation; Health Behavior; Eating behavior
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Body Weight Changes; Body Weight; Emotional Regulation; Health Behavior; Feeding Behavior | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Stress Reduction (MBSR) program (Experimental): Mindfulness Based Stress Reduction (MBSR) is an 8-week program that consists of training in mindfulness practices, the application of mindfulness to daily life, and information about healthy living and the role played by thoughts and emotions in health.
  Interventions: Behavioral: Mindfulness
- Healthy Living Course (HLC) (Active Comparator): Healthy Living Course (HLC) an 8-week psycho-educational program that consists of lectures and discussion on healthy living, stress management, time management, and unhealthy behaviors (e.g. smoking, drinking).
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness
  Arms: Mindfulness Based Stress Reduction (MBSR) program
Behavioral: Psychoeducation
  Arms: Healthy Living Course (HLC)

SUMMARY:
The goal of this project is to characterize changes in emotion regulation pathways associated with healthy behaviors in people who have recently lost weight and are seeking to maintain weight loss over a 1-year period.

DETAILED DESCRIPTION:
Unhealthy behaviors such as overeating and a sedentary lifestyle are largely responsible for overweight and obesity which substantially increase risk for chronic conditions such as heart disease, high blood pressure, stroke, diabetes, arthritis and certain cancers. The rapid rise in obesity threatens to reverse recent gains in life expectancy and account for a large percentage of premature deaths in the U.S. Although there is evidence for the short-term efficacy of a number of methods for initiating health behavior change to lose weight, these interventions have shown only limited ability to affect significant, long-term behavioral changes in the majority of adults. In part this may be because they fail to adequately address how psychological factors that lead to relapse to unhealthy behaviors and failure to maintain long-term behavior change.

The purpose of the study is to understand brain changes that accompany participation in programs that foster healthy behaviors in people seeking to maintain weight loss. We will use MRI scans to study brain function in men and women 25-60 years old who have lost weight in the last year without surgery. Participants will be assigned to one of two programs to help them maintain weight loss and will be compensated for their time. Our goal is to gain a better understanding of the brain changes that lead to long-term success in keeping weight off, in the hope that this knowledge will assist in the development of improved treatments.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 60 years old
* Healthy individuals who have intentionally lost at least 5% of their body weight over the past year
* BMI >20.5 kg/m2 at study entry and >25 in past 2 years

Exclusion Criteria:

* Weight-loss surgery or medications
* Serious Psychiatric or medical conditions
* Substance abuse
* Ineligible for MRI
* Pregnant
* Eating disorder

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Functional connectivity on fMRI | 8 weeks
  Functional Magnetic Resonance Imaging (fMRI)

SECONDARY OUTCOMES:
Association of functional connectivity change with changes in depression symptoms | 6 months
  Center for Epidemiological Studies-Depression Scale (CES-D)
Association of functional connectivity with maintenance of weight loss | 6 months
  BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Umass Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Fulwiler C, Siegel JA, Allison J, Rosal MC, Brewer J, King JA. Keeping Weight Off: study protocol of an RCT to investigate brain changes associated with mindfulness-based stress reduction. BMJ Open. 2016 Nov 30;6(11):e012573. doi: 10.1136/bmjopen-2016-012573. PMID 27903561